CLINICAL TRIAL: NCT00315224
Title: The Impact of Pulse Pressure on Cardiovascular Effects of Exercise Training in Hypertension of the Elderly
Brief Title: Sports in Hypertension of the Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EA4/019/2004
Record Dates: First submitted 2006-04-14; First posted 2006-04-18 (Estimated); Last update posted 2006-04-18 (Estimated); Status verified 2005-03

CONDITIONS: Hypertension
Keywords: Isolated systolic Hypertension; exercise; pulse pressure; endothelium
MeSH Terms: conditions — Hypertension; Isolated Systolic Hypertension; Motor Activity

INTERVENTIONS:
Behavioral: heart-rate controlled 12 week exercise program

SUMMARY:
The present work examines the impact of pulse pressure as a footprint of vascular ageing on cardiovascular benefits of endurance training in elderly hypertensives. METHODS AND RESULTS: 54 patients ≥ 60 years with antihypertensive treatment and diastolic 24h-ambulatory blood pressure (ABP) ≤ 90 mmHg are randomly assigned to sedentary activity or a heart-rate controlled 12 week exercise program, consisting of walking on a treadmill at target lactate concentrations of 2.5 ± 0.5 mmol/l. 24h-ambulatory blood pressure, physical performance, arterial elasticity, endothelium-derived vasodilation, quality of life, and weight are assessed at baseline and follow-up.

DETAILED DESCRIPTION:
Based on previous studies on sports in hypertension, we expected the intervention to result in a decrease of systolic 24h-ambulatory BP (systolic ABP) of at least 6 mm Hg in the training group with no changes in the control group.16,17 This difference was considered to be clinically relevant. A sample size of 23 in each group has 80% power to detect a difference in means of 6 mmHg assuming that the common standard deviation is 7 mmHg, a baseline systolic ABP of 140 mmHg and a two-sided p<0.05. We estimated the drop-out rate to be about 15% leading to a sample size of 27 patients per group.

Patients are recruited from our hypertension outpatient clinic. Inclusion criteria are current antihypertensive treatment, diastolic ABP ≤ 90 mmHg, age of ≥ 60 years. Prior to the exercise program, cardiac function is examined by ECG and echocardiogram. Exclusion criteria are regular engagement in physical exercise training in the past 12 weeks prior to inclusion in the study, symptomatic peripheral arterial occlusive disease, aortic insufficiency or stenosis > stage I, hypertrophic obstructive cardiomyopathy (HOCM), congestive heart failure (> NYHA II), uncontrolled cardiac arrhythmia with haemodynamic relevance, systolic office BP ≥ 180 mmHg, signs of acute ischemia in exercise ECG, change of antihypertensive medication in the past 6 weeks prior to inclusion in the study or during follow-up period. According to these criteria 54 patients are enrolled and randomized to exercise and control group.

Physical performance is assessed using a modified Bruce-protocol. Arterial elasticity is measured by pulse-wave analysis of the radial artery. Endothelium-dependent vasodilation is assessed sonographically by flow-mediated vasodilation. 24h-ABP monitoring is performed using Spacelabs 90207 monitors. The follow-up BP and vascular measurements of the training group are conducted within 2 days after the last training session.

The training program, consisting of walking on a treadmill according to an interval-training pattern, is carried out 3 times weekly for 12 weeks. If patients miss a training session, the program is prolonged until 36 workouts are carried out. The initial duration of training sessions is 30 minutes. During the first week, training consists of 5 workloads of 3 min; between workloads patients walk with half-speed for 3 min. Exercise duration is gradually increased to 4 x 5 min a day in the second week, 3 x 8 min in the third, 3 x 10 min in the fourth and 2 x 15 min in the fifth week. In the sixth and further weeks, exercise is progressively increased to 30, 32 and 36 min and is carried out without interruption. Training intensity corresponds to the speed necessary to reach a lactate concentration of 2.5 ± 0.5 mmol/l in capillary blood slightly above the aerobic threshold. Heart rate during training is controlled by a heart-rate monitor. As lactate concentration sinks below 2.0 mmol/l or exercise heart rate decreases by more than 5/min as a result of training adaptation, treadmill speed is increased by 0.5 km/h or elevation is increased by 3% to maintain training intensity. We have previously shown that this training protocol leads to a substantial increase of physical performance in short time. During training patients are continuously supervised by a physician.

ELIGIBILITY:
Inclusion Criteria:

≥ 60 years antihypertensive treatment diastolic 24h-ambulatory blood pressure (ABP) ≤ 90 mmHg

Exclusion Criteria:

regular engagement in physical exercise training in the past 12 weeks symptomatic peripheral arterial occlusive disease aortic insufficiency or stenosis > stage I hypertrophic obstructive cardiomyopathy (HOCM) congestive heart failure (> NYHA II) uncontrolled cardiac arrhythmia with haemodynamic relevance systolic office BP ≥ 180 mmHg signs of acute ischemia in exercise ECG change of antihypertensive medication in the past 6 weeks or during follow-up period

Min Age: 61 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54
Dates: Start 2005-02; Study Completion 2005-10

PRIMARY OUTCOMES:
Decrease of 24h-ambulatory systolic blood pressure

SECONDARY OUTCOMES:
change of diastolic blood pressure
change of pulse pressure
change of arterial compliance
change of endothelium-derived vasodilation

CONTACTS AND LOCATIONS:
Overall Officials: Timm H Westhoff, MD, Principal Investigator — Charité, Campus Benjamin Franklin, Medizinische Klinik IV, Berlin, Germany
Locations (1):
- Charité, Campus Benjamin Franklin, Berlin, Germany